CLINICAL TRIAL: NCT06660784
Title: Mechanism of Nitric Oxide on Ventilator-induced Diaphragm Dysfunction with Extracorporeal Membrane Lung Assistance
Status: Active, not recruiting | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PTXM2024028
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-09

CONDITIONS: Tracheal Intubation; Extracorporeal Membrane Oxygenation; Nitric Oxide; Ventilator-induced Diaphragmatic Dysfunction
Keywords: ventilator-induced diaphragm dysfunction; nitric oxide; extracorporeal membrane oxygenation; oxidative stress; endoplasmic reticulum stress
MeSH Terms: interventions — Nitric Oxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Nitric Oxide — Depending on the indication, the subjects will be given NO treatment or not. In ECMO assisted mechanical ventilation + NO treatment group, the subjects will be randomly assigned to NO treatment via ventilator or membrane oxygenator.

SUMMARY:
The goal of this clinical trial is to explore the effect of NO treatment on diaphragm function after mechanical ventilation with ECMO assistance. We expect to enroll a total of 80 patients who will receive mechanical ventilation and mechanical ventilation combined with ECMO treatment. Depending on the indication, they will be given NO treatment or not. In ECMO assisted mechanical ventilation + NO treatment group, the subjects will be randomly assigned to NO treatment via ventilator or membrane oxygenator. The main questions it aims to answer are:

1. Observing the influences and potential therapeutic effects of different NO insertion methods through ventilator or membrane oxygenator on the occurrence and development of ventilator-induced diaphragm (VIDD) dysfunction during ECMO assisted mechanical ventilation.
2. Exploring the potential key molecular mechanisms of NO treatment on the occurrence and development of VIDD after ECMO assisted mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Tracheal intubation in our emergency department;
3. Expected survival time ≥ 72 hours;
4. Family members agree to participate and sign the informed consent form.

Exclusion Criteria:

1. Pregnant women;
2. Patients with diaphragmatic hernia or other known diaphragmatic diseases and injuries;
3. Patients with mechanical ventilation treatment within 3 months;
4. Thoracic or abdominal tumor invading the diaphragm;
5. A large amount of ascites raises the diaphragm position;
6. Upper respiratory tract malformation;
7. Trauma leading to chest collapse, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of mechanical ventilation with or without ECMO assistance in emergency ward
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Diaphragm function | We starts POCUS within 1 hour (1h) after mechanical ventilation, and continuously monitoring the diaphragm function at 6h, 12h, 24h, 48h, 72h, 96h, 120h, 144h and 168h respectively. POCUS will be terminated if the patient dies.
  Continuous POCUS monitoring of diaphragm function during mechanical ventilation, including diaphragm thickness, diaphragm thickening fraction, diaphragm excursion, etc

SECONDARY OUTCOMES:
Inflammatory cytokines | The fixed time point on the 1st, 2nd, 3rd, 4th, 5th, 6th and 7th day.
  TNF - α, IL-1β , IL-6, IL-8, IL-10, etc.
Oxidative stress markers | The fixed time point on the 1st, 2nd, 3rd, 4th, 5th, 6th and 7th day.
  ROS, SOD, MDA, GSH, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hetz C. The unfolded protein response: controlling cell fate decisions under ER stress and beyond. Nat Rev Mol Cell Biol. 2012 Jan 18;13(2):89-102. doi: 10.1038/nrm3270. PMID 22251901
- [Background] Jiao G, Hao L, Wang M, Zhong B, Yu M, Zhao S, Wang P, Feng R, Tan S, Chen L. Upregulation of endoplasmic reticulum stress is associated with diaphragm contractile dysfunction in a rat model of sepsis. Mol Med Rep. 2017 Jan;15(1):366-374. doi: 10.3892/mmr.2016.6014. Epub 2016 Dec 9. PMID 27959404
- [Background] Maes K, Stamiris A, Thomas D, Cielen N, Smuder A, Powers SK, Leite FS, Hermans G, Decramer M, Hussain SN, Gayan-Ramirez G. Effects of controlled mechanical ventilation on sepsis-induced diaphragm dysfunction in rats. Crit Care Med. 2014 Dec;42(12):e772-82. doi: 10.1097/CCM.0000000000000685. PMID 25402297
- [Background] Liu YY, Li LF. Ventilator-induced diaphragm dysfunction in critical illness. Exp Biol Med (Maywood). 2018 Dec;243(17-18):1329-1337. doi: 10.1177/1535370218811950. Epub 2018 Nov 19. PMID 30453774
- [Background] Gallot YS, Bohnert KR. Confounding Roles of ER Stress and the Unfolded Protein Response in Skeletal Muscle Atrophy. Int J Mol Sci. 2021 Mar 4;22(5):2567. doi: 10.3390/ijms22052567. PMID 33806433
- [Background] Bohnert KR, McMillan JD, Kumar A. Emerging roles of ER stress and unfolded protein response pathways in skeletal muscle health and disease. J Cell Physiol. 2018 Jan;233(1):67-78. doi: 10.1002/jcp.25852. Epub 2017 May 16. PMID 28177127
- [Background] Afroze D, Kumar A. ER stress in skeletal muscle remodeling and myopathies. FEBS J. 2019 Jan;286(2):379-398. doi: 10.1111/febs.14358. Epub 2017 Dec 29. PMID 29239106
- [Background] Shen J, Prywes R. Dependence of site-2 protease cleavage of ATF6 on prior site-1 protease digestion is determined by the size of the luminal domain of ATF6. J Biol Chem. 2004 Oct 8;279(41):43046-51. doi: 10.1074/jbc.M408466200. Epub 2004 Aug 6. PMID 15299016
- [Background] Yoshida H, Matsui T, Yamamoto A, Okada T, Mori K. XBP1 mRNA is induced by ATF6 and spliced by IRE1 in response to ER stress to produce a highly active transcription factor. Cell. 2001 Dec 28;107(7):881-91. doi: 10.1016/s0092-8674(01)00611-0. PMID 11779464
- [Background] Haze K, Yoshida H, Yanagi H, Yura T, Mori K. Mammalian transcription factor ATF6 is synthesized as a transmembrane protein and activated by proteolysis in response to endoplasmic reticulum stress. Mol Biol Cell. 1999 Nov;10(11):3787-99. doi: 10.1091/mbc.10.11.3787. PMID 10564271
- [Background] Oida Y, Shimazawa M, Imaizumi K, Hara H. Involvement of endoplasmic reticulum stress in the neuronal death induced by transient forebrain ischemia in gerbil. Neuroscience. 2008 Jan 2;151(1):111-9. doi: 10.1016/j.neuroscience.2007.10.047. Epub 2007 Nov 13. PMID 18082969
- [Background] Tajiri S, Oyadomari S, Yano S, Morioka M, Gotoh T, Hamada JI, Ushio Y, Mori M. Ischemia-induced neuronal cell death is mediated by the endoplasmic reticulum stress pathway involving CHOP. Cell Death Differ. 2004 Apr;11(4):403-15. doi: 10.1038/sj.cdd.4401365. PMID 14752508
- [Background] Mamady H, Storey KB. Coping with the stress: expression of ATF4, ATF6, and downstream targets in organs of hibernating ground squirrels. Arch Biochem Biophys. 2008 Sep 1;477(1):77-85. doi: 10.1016/j.abb.2008.05.006. Epub 2008 May 25. PMID 18541136
- [Background] Vattem KM, Wek RC. Reinitiation involving upstream ORFs regulates ATF4 mRNA translation in mammalian cells. Proc Natl Acad Sci U S A. 2004 Aug 3;101(31):11269-74. doi: 10.1073/pnas.0400541101. Epub 2004 Jul 26. PMID 15277680
- [Background] Wek RC, Jiang HY, Anthony TG. Coping with stress: eIF2 kinases and translational control. Biochem Soc Trans. 2006 Feb;34(Pt 1):7-11. doi: 10.1042/BST20060007. PMID 16246168
- [Background] Harding HP, Zhang Y, Ron D. Protein translation and folding are coupled by an endoplasmic-reticulum-resident kinase. Nature. 1999 Jan 21;397(6716):271-4. doi: 10.1038/16729. PMID 9930704
- [Background] Bommiasamy H, Popko B. Animal models in the study of the unfolded protein response. Methods Enzymol. 2011;491:91-109. doi: 10.1016/B978-0-12-385928-0.00006-7. PMID 21329796
- [Background] Ashraf NU, Sheikh TA. Endoplasmic reticulum stress and Oxidative stress in the pathogenesis of Non-alcoholic fatty liver disease. Free Radic Res. 2015;49(12):1405-18. doi: 10.3109/10715762.2015.1078461. Epub 2015 Aug 25. PMID 26223319
- [Background] Coggan AR, Peterson LR. Dietary Nitrate Enhances the Contractile Properties of Human Skeletal Muscle. Exerc Sport Sci Rev. 2018 Oct;46(4):254-261. doi: 10.1249/JES.0000000000000167. PMID 30001275
- [Background] Colussi C, Mozzetta C, Gurtner A, Illi B, Rosati J, Straino S, Ragone G, Pescatori M, Zaccagnini G, Antonini A, Minetti G, Martelli F, Piaggio G, Gallinari P, Steinkuhler C, Clementi E, Dell'Aversana C, Altucci L, Mai A, Capogrossi MC, Puri PL, Gaetano C. HDAC2 blockade by nitric oxide and histone deacetylase inhibitors reveals a common target in Duchenne muscular dystrophy treatment. Proc Natl Acad Sci U S A. 2008 Dec 9;105(49):19183-7. doi: 10.1073/pnas.0805514105. Epub 2008 Dec 1. PMID 19047631
- [Background] Hu RG, Sheng J, Qi X, Xu Z, Takahashi TT, Varshavsky A. The N-end rule pathway as a nitric oxide sensor controlling the levels of multiple regulators. Nature. 2005 Oct 13;437(7061):981-6. doi: 10.1038/nature04027. PMID 16222293
- [Background] Rassier DE, Kashina A. Protein arginylation of cytoskeletal proteins in the muscle: modifications modifying function. Am J Physiol Cell Physiol. 2019 May 1;316(5):C668-C677. doi: 10.1152/ajpcell.00500.2018. Epub 2019 Feb 21. PMID 30789755
- [Background] Cornachione AS, Leite FS, Wang J, Leu NA, Kalganov A, Volgin D, Han X, Xu T, Cheng YS, Yates JR 3rd, Rassier DE, Kashina A. Arginylation of myosin heavy chain regulates skeletal muscle strength. Cell Rep. 2014 Jul 24;8(2):470-6. doi: 10.1016/j.celrep.2014.06.019. Epub 2014 Jul 10. PMID 25017061
- [Background] Gupta MP, Samant SA, Smith SH, Shroff SG. HDAC4 and PCAF bind to cardiac sarcomeres and play a role in regulating myofilament contractile activity. J Biol Chem. 2008 Apr 11;283(15):10135-46. doi: 10.1074/jbc.M710277200. Epub 2008 Feb 4. PMID 18250163
- [Background] Lundberg JO, Weitzberg E, Gladwin MT. The nitrate-nitrite-nitric oxide pathway in physiology and therapeutics. Nat Rev Drug Discov. 2008 Feb;7(2):156-67. doi: 10.1038/nrd2466. PMID 18167491
- [Background] Lundberg JO, Govoni M. Inorganic nitrate is a possible source for systemic generation of nitric oxide. Free Radic Biol Med. 2004 Aug 1;37(3):395-400. doi: 10.1016/j.freeradbiomed.2004.04.027. PMID 15223073
- [Background] Kobzik L, Reid MB, Bredt DS, Stamler JS. Nitric oxide in skeletal muscle. Nature. 1994 Dec 8;372(6506):546-8. doi: 10.1038/372546a0. PMID 7527495
- [Background] Stamler JS, Meissner G. Physiology of nitric oxide in skeletal muscle. Physiol Rev. 2001 Jan;81(1):209-237. doi: 10.1152/physrev.2001.81.1.209. PMID 11152758
- [Background] Malfertheiner MV, Garrett A, Passmore M, Haymet AB, Webb RI, Von Bahr V, Millar JE, Schneider BA, Obonyo NG, Black D, Bouquet M, Bartnikowski N, Suen JY, Fraser JF. The effects of nitric oxide on coagulation and inflammation in ex vivo models of extracorporeal membrane oxygenation and cardiopulmonary bypass. Artif Organs. 2023 Oct;47(10):1581-1591. doi: 10.1111/aor.14608. Epub 2023 Jul 19. PMID 37395735
- [Background] Toomasian JM, Jeakle MMP, Langley MW, Poling CJ, Lautner G, Lautner-Csorba O, Meyerhoff MM, Carr BJD, Rojas-Pena A, Haft JW, Bartlett RH. Nitric Oxide Attenuates the Inflammatory Effects of Air During Extracorporeal Circulation. ASAIO J. 2020 Jul;66(7):818-824. doi: 10.1097/MAT.0000000000001057. PMID 31425266
- [Background] Ciampa AR, de Prati AC, Amelio E, Cavalieri E, Persichini T, Colasanti M, Musci G, Marlinghaus E, Suzuki H, Mariotto S. Nitric oxide mediates anti-inflammatory action of extracorporeal shock waves. FEBS Lett. 2005 Dec 19;579(30):6839-45. doi: 10.1016/j.febslet.2005.11.023. Epub 2005 Nov 28. PMID 16325181
- [Background] Lahtinen M, Melki V, Adamik B, Khamis H, Borowiec JW. Nitric oxide and inflammatory response in simulated extracorporeal circulation. Thorac Cardiovasc Surg. 2003 Jun;51(3):130-7. doi: 10.1055/s-2003-40318. PMID 12833201
- [Background] Pichugin VV, Domnin SE, Sandalkin EV, Fedorov SA, Bober VV, Zhurko SA. Nitrogen Oxide-Added Extracorporeal Membrane Oxygenation for Treating Critical Acute Heart Failure after Cardiac Surgery. Sovrem Tekhnologii Med. 2021;13(4):57-62. doi: 10.17691/stm2021.13.4.06. Epub 2021 Aug 28. PMID 34603764
- [Background] Psotova H, Ostadal P, Mlcek M, Kruger A, Janotka M, Vondrakova D, Svoboda T, Hrachovina M, Taborsky L, Dudkova V, Strunina S, Kittnar O, Neuzil P. Ischemic Postconditioning and Nitric Oxide Administration Failed to Confer Protective Effects in a Porcine Model of Extracorporeal Cardiopulmonary Resuscitation. Artif Organs. 2016 Apr;40(4):353-9. doi: 10.1111/aor.12556. Epub 2015 Sep 28. PMID 26412075
- [Background] Moury PH, Zunarelli R, Bailly S, Durand Z, Behouche A, Garein M, Durand M, Verges S, Albaladejo P. Diaphragm Thickening During Venoarterial Extracorporeal Membrane Oxygenation Weaning: An Observational Prospective Study. J Cardiothorac Vasc Anesth. 2021 Jul;35(7):1981-1988. doi: 10.1053/j.jvca.2020.10.047. Epub 2020 Oct 29. PMID 33218955
- [Background] McDonald CI, Fraser JF, Coombes JS, Fung YL. Oxidative stress during extracorporeal circulation. Eur J Cardiothorac Surg. 2014 Dec;46(6):937-43. doi: 10.1093/ejcts/ezt637. Epub 2014 Jan 30. PMID 24482384
- [Background] Kumar R, Coggan AR, Ferreira LF. Nitric oxide and skeletal muscle contractile function. Nitric Oxide. 2022 May 1;122-123:54-61. doi: 10.1016/j.niox.2022.04.001. Epub 2022 Apr 8. PMID 35405336
- [Background] van den Berg M, Hooijman PE, Beishuizen A, de Waard MC, Paul MA, Hartemink KJ, van Hees HWH, Lawlor MW, Brocca L, Bottinelli R, Pellegrino MA, Stienen GJM, Heunks LMA, Wust RCI, Ottenheijm CAC. Diaphragm Atrophy and Weakness in the Absence of Mitochondrial Dysfunction in the Critically Ill. Am J Respir Crit Care Med. 2017 Dec 15;196(12):1544-1558. doi: 10.1164/rccm.201703-0501OC. PMID 28787181
- [Background] Zhou XL, Wei XJ, Li SP, Liu RN, Yu MX, Zhao Y. Interactions between Cytosolic Phospholipase A2 Activation and Mitochondrial Reactive Oxygen Species Production in the Development of Ventilator-Induced Diaphragm Dysfunction. Oxid Med Cell Longev. 2019 Apr 18;2019:2561929. doi: 10.1155/2019/2561929. eCollection 2019. PMID 31178955
- [Background] Azuelos I, Jung B, Picard M, Liang F, Li T, Lemaire C, Giordano C, Hussain S, Petrof BJ. Relationship between Autophagy and Ventilator-induced Diaphragmatic Dysfunction. Anesthesiology. 2015 Jun;122(6):1349-61. doi: 10.1097/ALN.0000000000000656. PMID 25828754
- [Background] Karagiannidis C, Lubnow M, Philipp A, Riegger GA, Schmid C, Pfeifer M, Mueller T. Autoregulation of ventilation with neurally adjusted ventilatory assist on extracorporeal lung support. Intensive Care Med. 2010 Dec;36(12):2038-44. doi: 10.1007/s00134-010-1982-6. Epub 2010 Aug 6. PMID 20689930
- [Background] Riccardo Pinciroli, Alfio Bronco, Alberto Lucchini, and Giuseppe Foti.Acute Respiratory Failure: Ventilatory Support and Extracorporeal Membrane Oxygenation (ECMO).Springer International Publishing AG, part of Springer Nature.2019;51:733-748.
- [Background] Doorduin J, Roesthuis LH, Jansen D, van der Hoeven JG, van Hees HWH, Heunks LMA. Respiratory Muscle Effort during Expiration in Successful and Failed Weaning from Mechanical Ventilation. Anesthesiology. 2018 Sep;129(3):490-501. doi: 10.1097/ALN.0000000000002256. PMID 29771711
- [Background] Watson AC, Hughes PD, Louise Harris M, Hart N, Ware RJ, Wendon J, Green M, Moxham J. Measurement of twitch transdiaphragmatic, esophageal, and endotracheal tube pressure with bilateral anterolateral magnetic phrenic nerve stimulation in patients in the intensive care unit. Crit Care Med. 2001 Jul;29(7):1325-31. doi: 10.1097/00003246-200107000-00005. PMID 11445679